CLINICAL TRIAL: NCT01163058
Title: Retrospective Analysis Evaluating Molecular Factors of Primary Resistance to Tyrosine Kinase Inhibitors in Metastatic Non Small Cell Lung Cancer Patients
Brief Title: Tyrosine Kinase Inhibitors In Metastatic Non Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Armando Santoro, MD, Istituto Clinico Humanitas
Other Study IDs: ONC/OSS-01/2010
Record Dates: First submitted 2010-06-29; First posted 2010-07-15 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim of the present retrospective study is to evaluate molecular factors of primary resistance to tyrosine kinase inhibitors in metastatic non small cell lung cancer (NSCLC) patients. The investigators assess first, the incidence of epidermal growth factor receptor (EGFR) and Kirsten ras sarcoma viral oncogene homolog (KRAS) mutations, SOS and hepatocyte growth factor (HGF) expression, anaplastic lymphoma kinase (ALK) translocation and expression and, secondly, the investigators correlate molecular markers with clinical features and outcome in terms of response rate, progression free survival and overall survival.

DETAILED DESCRIPTION:
Non small cell lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of NSCLC (non small cell lung cancer) with available tumor tissue for mutational analysis
* Metastatic disease treated with gefitinib or erlotinib
* Presence of at least one measurable lesion according to RECIST criteria

Exclusion Criteria:

* No tumor tissue available
* No clinical data available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non small cell lung cancer patients treated with gefitinib or erlotinib
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Determine the incidence of EGFR (Epidermal growth factor ) and KRAS (Kirsten ras sarcoma viral oncogene homolog ) mutations in 300 NSCLC (non small cell lung cancer) patients treated with gefitinib or erlotinib | 1 year

SECONDARY OUTCOMES:
Investigate the association of clinical features such as sex, age, smoking history and histology with oncogenic alterations. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy